CLINICAL TRIAL: NCT01974973
Title: Open Label Study of Autologous Bone Marrow Mononuclear Cells in Autism Spectrum Disorders
Brief Title: Stem Cell Therapy in Autism Spectrum Disorders
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-02
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorders
Keywords: autism spectrum disorders; stem cells
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cell (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Procedure: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Procedure: Autologous bone marrow mononuclear cell transplantation — Intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to study the effect of stem cell therapy on common symptoms in patients with autism spectrum disorders

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of any type of autism spectrum disorders
* age above 6 months

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Improvement in the scales for Autism spectrum disorders | Six months

SECONDARY OUTCOMES:
Positron Emission Tomography- computed tomography to study change in brain metabolism | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geffner LF, Santacruz P, Izurieta M, Flor L, Maldonado B, Auad AH, Montenegro X, Gonzalez R, Silva F. Administration of autologous bone marrow stem cells into spinal cord injury patients via multiple routes is safe and improves their quality of life: comprehensive case studies. Cell Transplant. 2008;17(12):1277-93. doi: 10.3727/096368908787648074. PMID 19364066